CLINICAL TRIAL: NCT05032677
Title: Comparative Study Between Dural Puncture Epidural Technique Versus Conventional Epidural Technique During Laparoscopic Hysterectomy
Brief Title: Dural Puncture Epidural Technique Versus Conventional Epidural Techmique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Ali Abdelhaleem Abdelrahman, Anesthesia lecturer M.D., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ES-2022
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Gynecologic Disease Requiring Laparoscopic Hysterectomy Under Neuraxial Anesthesia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Epidural Technique (Experimental)
  Interventions: Procedure: Dural Puncture Epidural Technique using pencil-point 25G Whitacre needle
- Dural Puncture Epidural technique using pencil-point 25G Whitacre needle (Active Comparator)
  Interventions: Procedure: Conventional Epidural Technique

INTERVENTIONS:
Procedure: Conventional Epidural Technique — Standard Lumbar Epidural Block using Touhy Epidural Needle (18G) at L2-3 inter-space and Epidural Catheter (20G) was inserted then bupivacaine 0.5% 15-20 ml with 50ug fentanyl was given.
  Arms: Dural Puncture Epidural technique using pencil-point 25G Whitacre needle
Procedure: Dural Puncture Epidural Technique using pencil-point 25G Whitacre needle — 25G Dural Puncture Epidural Block at L2-3 inter-space then bupivacaine 0.5% 15-20 ml with 50ug fentanyl was given.
  Arms: Conventional Epidural Technique

SUMMARY:
This study will be conducted on 50 patients of ASA grade I and II aged from 25 to 55 years and presented for laparoscopic hysterectomy. Patients will be divided into two equal groups; group A control group for conventional epidural technique(n=25) and group B for 25G dural puncture epidural with 25G pencil point Whitacre spinal needle (n=25). Randomization will be done using computer generated number and concealed using sequentially numbered, sealed opaque envelope.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II
* Height(150-170 cm)

Exclusion Criteria:

* patient refusal
* hypersensitivity to local anesthetic drugs
* bleeding disorders and coagulopathy(platelets count less than 80000,INR less than 1.5 or therapeutic dose of anticoagulant).

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
incidence of bilateral sacral blockade | Up to 30 minutes after local anesthetic injection
  Sensory blockade was evaluated using a non-traumatic pinprick stimulus starting at the S2 dermatome and moving in a caudad direction (measured every 2 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Reham Ali Abdelrahman, M.D., Principal Investigator — Cairo University
Locations (1):
- Department of Anesthesia, Surgical ICU, and Pain Management, Cairo, Egypt